CLINICAL TRIAL: NCT05991219
Title: Screening and Secondary Prevention Rheumatic Heart Disease
Brief Title: Screening and Secondary Prevention Rheumatic Heart Disease Study
Acronym: S2-RHD
Status: Recruiting | Type: Observational
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Responsible Party: Principal Investigator, Sabha Bhatti, Professor, National Institute of Cardiovascular Diseases, Pakistan
Other Study IDs: IRB-32/2023
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Rheumatic Heart Disease
MeSH Terms: conditions — Rheumatic Heart Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
After basic clinical screening including history and physical, Point of care ultrasound will be performed to look at Mitral, Aortic and Tricuspid Valves for regurgitation or stenosis. For patients with confirmed Rheumatic heart disease (RHD), treatment and referral depending on stage of disease. Antibiotic prescription could be shifted to community health workers delivering preventive medications via practical clinical algorithms, diagnostic tools, availability of appropriate antibiotics, and supportive supervision. Patients will have repeat imaging at 2 years and 5 years to look at the outcome of delayed progression of valve disease.

DETAILED DESCRIPTION:
Screening for RHD should be carried out since it is a major health concern that has been shown to have a treatable and detectable latent stage that can be diagnosed using a simple sensitive test (point of care ultrasound) and early treatment (secondary prevention using antibiotic prophylaxis) can provide a better outcome (slow progression of disease) in a cost effective way. The investigators aim to study the Incidence and Prevalence of RHD in community and school settings and aim to intervene depending on the stage the disease is picked up in.

ELIGIBILITY:
Inclusion Criteria:

* Rural communities in Sindh

Exclusion Criteria:

* Refused to participate in the study

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Age group 10-30 years. Screening in rural communities in Sindh including very low income areas outside Karachi. Schools (free government schools in low income areas) and patient point of contact locations such as National Institute of Cardiovascular Diseases Pakistan Satellite centers (10) and chest pain units (24) will also be utilized. Family members of patients with known rheumatic heart disease will also be screened.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Rheumatic heart disease | At the time of screening echocardiogram
  Number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Sabha Bhatti, MD, Principal Investigator — National Institute of Cardiovascular Diseases
Locations (1):
- National Institute of Cardiovascular Diseases (NICVD), Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No